CLINICAL TRIAL: NCT00760045
Title: Clinical Pharmacological Study of AL-43546 Ophthalmic Product in Subjects With Shortened Tear Film Break Up Time
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Koji Hasegawa, Alcon
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: C-07-54
Record Dates: First submitted 2008-09-24; First posted 2008-09-25 (Estimated); Last update posted 2010-01-06 (Estimated); Status verified 2010-01

CONDITIONS: Dry Eye Disease
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): AL-43546 0.15%
  Interventions: Drug: Hydroxypropyl Guar Galactomannan
- 2 (Experimental): AL-43546 0.25%
  Interventions: Drug: Hydroxypropyl Guar Galactomannan
- 3 (Active Comparator): AL-43546 0%(Vehicle)
  Interventions: Drug: Hydroxypropyl Guar Galactomannan
- 4 (Active Comparator): 0.1% sodium hyaluronate ophthalmic solutio
  Interventions: Drug: 0.1% sodium hyaluronate ophthalmic solution

INTERVENTIONS:
Drug: Hydroxypropyl Guar Galactomannan — One drop per one time in both eyes, once daily (at each visit).One instillation daily in one period and a total of 4 instillations over 4 periods.
  Arms: 1; 2; 3
Drug: 0.1% sodium hyaluronate ophthalmic solution — One drop per one time in both eyes, once daily (at each visit).One instillation daily in one period and a total of 4 instillations over 4 periods.
  Arms: 4

SUMMARY:
The purpose of the study is to observe lacrimal fluid condition (tear film break-up time) chronologically after a single dose of AL-43546 ophthalmic products（0.15%, 0.25% and vehicle）and 0.1% sodium hyaluronate ophthalmic solution and compare lacrimal fluid retention time between them.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with NIBUT of either eye is 8 seconds or less and other eye is 10 seconds or less at screening test and NIBUT of either eye before instillation in Period I is 10 seconds or less.

Exclusion Criteria:

* Diagnosis of severe Sjogren's syndrome (history of the use of punctal plug one time or more, etc.) in either eye.
* Subjects who will use ophthalmic solutions (excluding the specified artificial tear) or ophthalmic ointment in either eye during the study period.

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2008-08; Primary Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
The change from baseline of non-invasive tear film break up time (ΔNIBUT: seconds). | Up to 180 minutes

SECONDARY OUTCOMES:
Ocular comfort | After installation

CONTACTS AND LOCATIONS:
Locations (1):
- Osaka Pharmacology Clinical Research Hospital, Osaka, Osaka, Japan